CLINICAL TRIAL: NCT06861010
Title: Evaluating the Safety and Efficacy of Ondansetron in the Prevention of Post Endoscopic Retrograde Cholangiopancreatography Pancreatitis
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mostafa Bahaa, Lecturer, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 54782
Record Dates: First submitted 2025-03-01; First posted 2025-03-06 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Pancreatic Diseases
MeSH Terms: conditions — Pancreatic Diseases | interventions — Ondansetron

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: double blinded
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Placebo Comparator): the patients will receive placebo tablet 2 h before ERCP
  Interventions: Other: Placebo
- ondansetron group (Active Comparator): the patients will receive placebo tablet 2 h before ERCP.
  Interventions: Drug: Ondansetron

INTERVENTIONS:
Other: Placebo — Placebo tablets will have the same look and appearance of ondansetron.
  Arms: Control group
Drug: Ondansetron — ondansetron is commonly used as anti-emetics to prevent and treat chemotherapy-induced vomiting and nausea
  Arms: ondansetron group

SUMMARY:
Endoscopic retrograde cholangiopancreatography (ERCP (, a key tool that is used in diagnosis and treatment of pancreato-biliary diseases. Post-ERCP pancreatitis (PEP) is the most common and serious complication that can occur following this procedure and can lead to significant morbidity and mortality. A variety of patient-related and procedure-related factors have been associated with higher rates of PEP.

ELIGIBILITY:
Inclusion Criteria:

1. Age more than 18 years old.
2. Gender: Males and Females
3. Patients with suitable indications for ERCP due to suspected pancreato-biliary disorders.
4. Blood amylase and lipase levels before ERCP are within the normal limits.

Exclusion Criteria:

1. Age of less than18 years.
2. Uncontrolled diabetes mellitus (DM)
3. Severe bleeding tendency
4. Impaired renal function (serum creatinine > 2 mg/dL), (creatinine clearance <30 ml/min)
5. Patients with severe heart disease.
6. Subjects who underwent prior biliary or pancreatic sphincterotomy or dilatation or stenting of either duct.
7. Currently pregnant or nursing
8. Admission due to established pancreatitis before ECRP
9. Unwillingness to undergo ERCP.
10. Previously documented allergy to ondansetron.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-12-20 (Estimated); Study Completion 2025-12-20 (Estimated)

PRIMARY OUTCOMES:
The primary outcome that will be measured is the development of pancreatitis after the procedure according to consensus criteria | 24 hours
  The primary outcome that will be measured is the development of pancreatitis after the procedure according to consensus criteria. Briefly in this criteria PEP will be diagnosed if the Patient met two of the three following criteria after ERCP: new onset or increased abdominal pain consistent with acute pancreatitis, pancreatic enzyme elevation to at least 3 times the upper limit of normal at 24 hours after the procedure, and the necessity for new or continued hospitalization for at least 2 nights

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta Unuversity, Tanta, Egypt